CLINICAL TRIAL: NCT01327482
Title: Modeling Intracellular and Extracellular Raltegravir (RAL) Pharmacokinetics in the Female Genital Tract and Blood After a Twice Daily 400mg Dose Over the Course of a Menstrual Cycle
Brief Title: Levels of Raltegravir in the Female Genital Tissue
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Caroline Mitchell, Assistant Professor, University of Washington
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 38681-D
Record Dates: First submitted 2011-03-30; First posted 2011-04-01 (Estimated); Results first posted 2014-12-19 (Estimated); Last update posted 2014-12-19 (Estimated); Status verified 2014-12

CONDITIONS: HIV
Keywords: Raltegravir; Pharmacokinetics
MeSH Terms: interventions — Raltegravir Potassium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- All (Experimental): All patients were part of the intervention arm, as this was a pharmacokinetic study. All women took Raltegravir 400mg orally, twice daily for 3 weeks.
  Interventions: Drug: Raltegravir

INTERVENTIONS:
Drug: Raltegravir — Dosage: 400mg/PO (by mouth) Frequency: Twice daily Duration: During course of menstrual cycle (28 days)
  Other Names: Isentress

SUMMARY:
This study is an investigation of the pharmacokinetics of raltegravir in the tissue of the female genital tract to determine if twice-daily dosing of 400mg achieves adequate drug levels to prevent viral integration of HIV-1. The study will also assess whether drug levels change in the tissue across the different phases of the menstrual cycle.

* Hypothesis #1: Twice daily dosing with raltegravir 400mg will result in intracellular concentrations that should be sufficient to suppress HIV-1 replication throughout the menstrual cycle.
* Hypothesis #2: Intracellular genital raltegravir peaks will be lower and troughs higher compared to extracellular concentrations in the plasma and PMBCs (peripheral blood mononuclear cells).
* Hypothesis #3: Intracellular raltegravir concentrations will be slightly lower during the luteal phase of the menstrual cycle due to cellular pumps such as p-glycoprotein, which are present in higher numbers during periods of high progesterone.

DETAILED DESCRIPTION:
HIV-1 is shed in genital secretions which increase the risk of transmission between sexual partners and from mother to infant. Antiretroviral medication taken prior to exposure to HIV-1 can prevent viral transmission from a mother to her infant. Raltegravir (RAL), by blocking integration of viral cDNA into the host's genome, makes an excellent candidate for preventing HIV-1 infection. RAL is licensed for treatment with twice-daily dosing based on plasma trough concentrations; however, intracellular concentrations of RAL which are relevant to blocking infection of cells have not been previously studied. P-glycoprotein pumps, which are involved in regulating drug absorption and metabolism, can influence intracellular drug concentrations. P-glycoprotein concentrations appear to vary with menstrual cycle suggesting it may affect intracellular drug concentration of RAL in women.

Women will be enrolled in the study and followed during the course of a menstrual cycle while taking a dose of 400mg PO twice daily. An initial screening visit will be performed prior to enrollment and participation in the study. Review of medical history as well as blood and urine collection will occur during the screening visit. Once enrolled, participants will have blood and genital tract samples collected once a week for four weeks to assess intracellular concentrations of RAL in the blood and genital tract tissue.

ELIGIBILITY:
Inclusion Criteria

Volunteers must be:

* Over 18 years of age.
* Willing to abstain from sexual intercourse during course of study.
* Able to commit to follow-up visit schedule.
* Willing to abstain from use of vaginal medications or creams 48 hours prior to follow-up visits.
* Willing and able to provide informed consent.

Exclusion Criteria

Volunteers will not be eligible for the study if they:

* Are over 50 years of age.
* Are pregnant, attempting to become pregnant, or breast-feeding.
* Have irregular menstrual bleeding.
* Are using a hormonal form of birth control.
* Have abnormal liver/kidney function test results at screening visit.
* Have HIV-positive test result at screening visit.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2011-10; Primary Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Caroline Mitchell, MD, Principal Investigator — University Washington; Lisa Frenkel, MD, Principal Investigator — Seattle Children's Hospital
Locations (1):
- University of Washington, Clinical Research Center, Seattle, Washington, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Raltegravir: Healthy volunteers who had regular menses and were not on hormonal contraception
Period: Overall Study
Arm/Group | Raltegravir
Started | 10
Completed | 9 (The 10th participant completed 2/3 visits)
Not Completed | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Arm/Group | Raltegravir
Number analyzed (Participants) | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 30 (8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 10

OUTCOME MEASURES:

1. Primary Outcome: Tissue Raltegravir Concentrations
Description: Mean trough concentration from all three days. Tissue concentrations are measured from cervical biopsy homogenate using a mass-spectroscopy-based method.
Time Frame: 7, 14, 21 days
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Raltegravir
Number analyzed (Participants) | 10
ng/mL | 117 (229)

2. Secondary Outcome: Plasma Raltegravir Concentrations
Description: Mean trough concentration from all 3 days
Time Frame: 7, 14, 21 days
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Raltegravir
Number analyzed (Participants) | 10
ng/mL | 160 (394)

ADVERSE EVENTS:
Arm/Group | Raltegravir
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 4/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Raltegravir (N=10)
Nausea (Gastrointestinal disorders) | 2 (2)
Vomiting (Gastrointestinal disorders) | 1 (1)
Knee pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No